CLINICAL TRIAL: NCT04358055
Title: Open-label, Multicenter, Prospective Investigation to Evaluate the Clinical Safety and Effectiveness of WET® Gel, Containing Hydeal-D®, an Ester of Hyaluronic Acid, in the Treatment of Nasal Dryness
Brief Title: Investigation to Evaluate the Clinical Safety and Effectiveness of WET® Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: QQ23_19_01
Record Dates: First submitted 2020-03-02; First posted 2020-04-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Nose Dry Feeling of
Keywords: dryness; nasal; gel; hyaluronic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WET® gel (Experimental): At the screening/baseline visit (Visit 1, Day 1), eligible patients will be assigned to treatment with WET® gel, at the dose of 3-4 nasal applications/day (according to necessity), 1or 2 puff/nostril, for maximum 14 days.
  Treatment will be administered according to patient's need without any relation with the time of the day (i.e. day time or night time administration), however within a maximum of 4 applications/day, which must include one administration in the morning upon awakening and one administration in the evening before retiring to bed.
  Interventions: Device: WET® gel

INTERVENTIONS:
Device: WET® gel — In each application, a puff should be administered in each nostril every two seconds, with minimal inspirations, up to a sensation of lubrication in the external conduct is perceived. Then the patient should proceed with short inspirations and light touching of ala of the nose, to favour the distribution of the gel. A maximum of 4 erogations (2/nostril) is allowed in each application session.
  Other Names: WET® gel, containing Hydeal-D®, an ester of hyaluronic acid

SUMMARY:
The objective of the investigation is to assess the clinical safety and effectiveness of WET® gel in the treatment of nasal dryness, following maximum two weeks of treatment.

DETAILED DESCRIPTION:
The objective of the project is to perform a post marketing clinical study to confirm safety and clinical effectiveness of WET® gel in the treatment of nasal dryness.

This investigation will be carried out following the CE marking of the WET® gel device and is mainly intended to answer questions relating to clinical safety or performance (i.e. residual risks) of the device when used in accordance whit its approved labelling.

The study is also aimed at defining the optimal dose regimen of WET® gel.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having undergone the informed consent process and having signed an approved consent form;
2. Male and female outpatients, aged ≥ 18 years;
3. Patients with nasal dryness of moderate-severe intensity, defined as a score ≥ 4 in a 0-10 numeric rating scale (NRS), with or without superficial microlesions;
4. Patients with absence of nasal discharge;
5. Patients having not taken oral or intranasal decongestants, antihistamines (by any route), corticosteroids (by any route), intranasal anticholinergics, leukotriene inhibitors, mucolytics (by any route), sodium cromoglycate (by any route) in the 4 weeks preceding the screening/baseline visit and agree not to take them during the investigation;
6. Patients with a cooperative attitude and ability to be trained to use correctly the investigational medical device, to adhere to the dosing and visit schedules, and agree to record symptoms' severity scores and use of the investigational device in a daily diary;
7. If female of child-bearing potential, they must have a negative urine pregnancy test at the screening visit and use a reliable form of contraception for a least 1 month prior to Screening and throughout the investigation. Note: to be considered females of non-child-bearing potential, females must be surgically sterile or postmenopausal as documented in medical history for at least 1 year.

Exclusion Criteria:

1. Patients with atopic or non-atopic rhinosinusitis in active phase;
2. Patients with anatomical abnormalities of the nose (turbinate hypertrophy, septal deviation, polyps) that would interfere with nasal airflow;
3. Patients with a medical history of nasal or sinus surgery in the previous 12 months;
4. Patients with upper respiratory tract or sinus infection;
5. Patients with rhinitis medicamentosa;
6. Patients with epistaxis;
7. Patients having received treatment with oral or intranasal decongestants, anti-histamines (by any route), corticosteroids (by any route), intranasal anticholinergics, leukotriene inhibitors, mucolytics (by any route), sodium cromoglycate (by any route) in the 4 weeks preceding the screening/baseline visit;
8. Patients having received treatment with antibiotics (by any route) in the 4 weeks preceding the screening/baseline visit;
9. Patients currently undergoing a progressive course of immunotherapy(hyposensitization);
10. Patients having performed a sinus lavage in the 2 weeks preceding the screening/baseline visit;
11. Patients with known or suspected allergy, hypersensitivity or intolerance to hyaluronic acid and/or any other component of the investigational device;
12. Patients with presence of any of the following clinical conditions: active or quiescent tuberculosis infection of the respiratory tract, untreated fungal, bacterial, systemic viral infections or ocular herpes simplex;
13. Patients with presence of other serious gastrointestinal, renal, hepatic, pulmonary, cardiovascular, or neurological disease that could interfere with the outcome of the investigation or the patient's ability to comply with investigation requirements;
14. Patients who have been diagnosed of cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas);
15. Pregnant (positive urine test) or breastfeeding women, or planning to become pregnant during the investigation;
16. Patients with history of alcoholism or drug dependence;
17. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the investigation;
18. Patients who have used any investigational drug or device, or have participated in an investigational protocol in the past 3 months;
19. Patients who have been previously enrolled in this investigation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability of WET® gel | 15 days (the entire study duration)
  The primary objective of the investigation is to evaluate the general safety and local tolerability of WET® gel in the primary endpoint incidence of treatment-related treatment-emergent adverse events (TEAEs). Endpoint: Incidence of local and general treatment-related TEAEs during the entire investigation duration.

SECONDARY OUTCOMES:
Change in nasal dryness | 15 days (the entire study duration)
  Changes from baseline in score (0-10 NRS) of nasal dryness (morning, evening and daily mean) at any post-baseline time points
Percentage of patients with resolution of nasal dryness | 15 days (the entire study duration)
  Percentage of patients with resolution of nasal dryness (defined as a score of 0 in the NRS for ≥ 3 consecutive days)
Time to resolution of nasal dryness | 15 days (the entire study duration)
  Time to resolution of nasal dryness (defined as a score of 0 in the NRS for ≥ 3 consecutive days)
Changes from baseline of nasal crusting | 15 days (the entire study duration)
  Changes from baseline in score (0-10 NRS) of nasal crusting (morning, evening and daily mean) at any post-baseline time point
Changes from baseline of nasal itching | 15 days (the entire study duration)
  Changes from baseline in score (0-10 NRS) of nasal itching (morning, evening and daily mean) at any post-baseline time point
Changes from baseline of nasal burning | 15 days (the entire study duration)
  Changes from baseline in score (0-10 NRS) of nasal burning (morning, evening and daily mean) at any post-baseline time point
Changes from baseline of nasal obstruction | 15 days (the entire study duration)
  Changes from baseline in score (0-10 NRS) of nasal obstruction (morning, evening and daily mean) at any post-baseline time point
Compliance to treatment with WET® gel | 15 days (the entire study duration)
  Compliance to treatment according to patient diary

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Giordan, Study Director — Fidia Farmaceutici s.p.a.
Locations (4):
- Italy (4):
  - ATS Insubria, Como, Via Varese 11
  - ATS Insubria, Alzate Brianza
  - ATS Insubria, Erba
  - ATS Insubria, Porlezza

IPD SHARING:
Plan to Share IPD: No